CLINICAL TRIAL: NCT07026604
Title: A Study on the Safety and Preliminary Efficacy of the Anti-CD38 Monoclonal Antibody Daratumumab in the Treatment of Refractory Familial Cerebral Cavernous Malformations
Brief Title: Daratumumab for Familial Cerebral Cavernous Malformations: A Single-Arm Safety and Efficacy Study
Acronym: CCM-DS01
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCM-DS01
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cavernous Malformation, Cerebral
Keywords: cavernous malformation; CD38; Daratumumab; immunotherapy
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- intervention (Experimental): Participants receive intravenous daratumumab (16 mg/kg weekly for 8 weeks), diluted in 1000 mL (first dose) or 500 mL (subsequent doses) of saline, with infusion rates escalated stepwise from 50 to 200 mL/h under vital sign monitoring. Premedication (antihistamines/analgesics) is administered 30 minutes prior to each infusion to mitigate reactions. Weekly laboratory tests (hematology, liver/kidney function) and post-treatment MRI (3-month follow-up) assess safety and efficacy.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Participants receive intravenous daratumumab (16 mg/kg weekly for 8 weeks), diluted in 1000 mL (first dose) or 500 mL (subsequent doses) of saline, with infusion rates escalated stepwise from 50 to 200 mL/h under vital sign monitoring. Premedication (antihistamines/analgesics) is administered 30 minutes prior to each infusion to mitigate reactions.

SUMMARY:
Cerebral cavernous malformation (CCM) is a common vascular abnormality of the brain, affecting 0.1%-0.5% of people. It often causes recurrent brain hemorrhages, epilepsy, and neurological impairments, with surgery being the main treatment. However, surgery carries high risks for patients with multiple lesions or lesions in critical areas, and no effective pharmacological treatment is available. CCM is linked to mutations in genes like CCM1, CCM2, CCM3, or MAP3K3, which activate the MEK5-ERK5-KLF2/4 pathway, disrupting endothelial function. Immune cell infiltration, particularly plasma cells with high CD38 expression, suggests a role for humoral immunity in CCM. Depleting B cells in mouse models reduced lesions and hemorrhages, but broad B cell depletion is risky.

To find a safer treatment, researchers tested anti-CD38 monoclonal antibodies in mice, showing that targeting CD38 reduced CCM lesion formation. Given the success of CD38-targeted therapies like daratumumab in treating multiple myeloma, this study proposes evaluating daratumumab for CCM in a single-center trial with 10 adult patients to assess its safety and efficacy.

DETAILED DESCRIPTION:
Cerebral cavernous malformation (CCM) is a vascular anomaly occurring within the brain, with a prevalence of approximately 0.1%-0.5% in the general population, representing the most common vascular malformation of the central nervous system. CCM is the leading cause of recurrent intracerebral hemorrhage in adolescents and can also induce epilepsy, neurological deficits, and other related symptoms. Currently, the mainstay of treatment for CCM is surgical resection via craniotomy. However, for patients with multiple lesions or lesions located within the brainstem or eloquent brain regions, surgical intervention carries a significant risk of severe functional impairment or even mortality. At present, no effective pharmacological treatments are available for CCM.

Studies have demonstrated that endothelial cell mutations in genes CCM1, CCM2, CCM3, or MAP3K3 are key drivers of CCM pathogenesis. These pathogenic mutations activate the MEK5-ERK5-KLF2/4 signaling axis within endothelial cells, disrupting endothelial barrier function and coagulation regulation, thereby leading to lesion formation. Nevertheless, it has been recognized that, in addition to these genetic mutations, essential co-factors such as endothelial cell proliferation are also required for CCM initiation and progression.

Our previous research revealed that the CCM lesion microenvironment is characterized by substantial infiltration of immune cells, including myeloid cells and lymphocytes. Further analysis of the enriched cell types and their functions indicated the presence of a large number of specific plasma cells within CCM lesions, suggesting a role for activated humoral immunity in CCM pathogenesis. Gene expression profiling of these plasma cells revealed a marked expression of CD38.

To clarify the role of B cell-mediated humoral immunity in CCM development, we employed B cell-depleting antibodies in mouse models of CCM. Depletion of B cells resulted in a significant reduction in both lesion burden and associated hemorrhage. However, pan-B cell depletion is associated with broad immunosuppressive effects, potential adverse events, and lacks therapeutic precision, thereby limiting its clinical applicability.

To identify a more precise therapeutic target, we tested the efficacy of anti-CD38 monoclonal antibodies in two distinct mouse models of CCM. Our results demonstrated that targeting CD38 effectively inhibited CCM lesion formation and progression.

In recent years, CD38-targeted immunotherapies have been widely applied in the treatment of plasma cell malignancies and autoimmune diseases, exhibiting favorable safety profiles and sustained efficacy. Notably, in hematologic malignancies such as multiple myeloma (MM), CD38 monoclonal antibodies have become a cornerstone of first-line treatment. Daratumumab, an anti-CD38 monoclonal antibody, was the first CD38-targeted therapy approved for MM treatment and has significantly improved patient survival outcomes, demonstrating excellent safety and efficacy in clinical practice.

Based on these findings, we propose to explore the therapeutic potential of daratumumab, an anti-CD38 monoclonal antibody, for the treatment of CCM.This study is an open-label, single-arm, single-center clinical trial aimed at evaluating the safety and efficacy of the CD38 monoclonal antibody daratumumab in the treatment of familial cerebral cavernous malformations (CCM). Adult patients who meet the inclusion criteria will be enrolled, with an expected sample size of 10 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosed with familial cerebral cavernous malformation (familial CCM) (diagnosis requires at least one of the following: multiple CCMs or ≥2 family members with CCM);
* Presence of clinical symptoms or history of symptomatic events: intracerebral hemorrhage, stroke, permanent or transient neurological deficits, seizures, disability, or any other neurological symptoms associated with cavernous malformations;
* Deemed unsuitable for surgical resection by a physician;
* Able to provide written informed consent;
* Participant is willing and able to attend outpatient follow-up visits.

Exclusion Criteria:

* Stable familial CCM lesions not requiring intervention;
* Presence of metal implants or other contraindications to MRI;
* History of statin therapy within the past 6 months;
* History of beta-blocker therapy within the past 6 months;
* Laboratory abnormalities: absolute neutrophil count <1 × 10⁹/L, platelet count <100 × 10⁹/L, ALT >2.5× upper limit of normal (ULN), ALP >2.5× ULN, bilirubin >1.5× ULN, serum creatinine >2× ULN;
* Known HIV positivity, hepatitis B virus seropositivity (excluding passive immunity from vaccination or immunoglobulin therapy), defined as HBsAg-positive and/or anti-HBs and anti-HBc positive, or known hepatitis C virus positivity;
* Chronic or ongoing active infections requiring systemic treatment (e.g., chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis);
* Poorly controlled comorbidities, including chronic obstructive pulmonary disease (COPD), severe asthma, poorly controlled diabetes, renal and/or hepatic failure;
* Cardiovascular diseases, including unstable angina, acute myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA Class II), arrhythmias requiring treatment (excluding premature beats or minor conduction abnormalities), deep vein thrombosis (excluding stable muscular vein thrombosis as judged by the investigator), pulmonary embolism, or other severe thromboembolic events, or history of deep vein thrombosis, pulmonary embolism, or severe thromboembolic events within 6 months prior to enrollment with a risk of recurrence as assessed by the investigator;
* Participation in other interventional medical research or clinical trials within 4 weeks prior to screening (observational, natural history, or epidemiological studies without interventions are allowed);
* Known allergic reactions to infused protein products;
* Pregnancy (positive urine or serum pregnancy test in premenopausal women without documented surgical sterilization) or lactation;
* Any condition (e.g., substance abuse, alcohol dependence) that, in the investigator's opinion, may compromise the participant's compliance with study requirements;
* Participant or legal guardian unable to provide informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe infusion-related reactions (IRRs) | Up to 2 month
  Incidence of severe infusion-related reactions (IRRs) (defined as any adverse reaction directly caused by the injection procedure or drug administration, including fever, chills, hyperhidrosis, headache, bronchospasm, myalgia, arthralgia, hypotension, hypertension, etc., where the reaction persists without rapid resolution after symptomatic treatment and/or infusion interruption, recurs after initial improvement, or results in clinical consequences requiring hospitalization).
Change in total lesion volume on MRI during treatment | Up to 2 month
  Change in total lesion volume on MRI during treatment (specifically comparing post-treatment SWI [Susceptibility Weighted Imaging] sequence imaging with baseline imaging).

SECONDARY OUTCOMES:
Incidence of neutropenia during treatment | Up to 2 month
  Incidence of neutropenia during treatment (defined as absolute neutrophil count [ANC] <1 × 10⁹/L accompanied by a single temperature measurement >38.3°C or persistent temperature ≥38°C for over 1 hour).
Incidence of anemia during treatment | Up to 2 month
  Incidence of anemia during treatment (defined as hemoglobin [Hgb] below the lower limit of normal).
Incidence of cytokine release syndrome (CRS) during treatment | Up to 2 month
  Incidence of cytokine release syndrome (CRS) during treatment (defined as temperature ≥38°C not attributable to other causes, assessed according to the American Society for Transplantation and Cellular Therapy [ASTCT] consensus criteria).
Incidence of moderate IRRs | Up to 2 month
  Incidence of moderate IRRs (defined as adverse reactions directly caused by injection or drug administration that resolve rapidly after symptomatic treatment and/or infusion interruption).
Incidence of mild IRRs | Up to 2 month
  Incidence of mild IRRs (defined as transient adverse reactions directly caused by injection or drug administration, requiring no symptomatic treatment or infusion interruption).
Change in volume of the largest lesion | Up to 2 month
  Change in volume of the largest lesion identified on baseline MRI during treatment.
Change in number of lesions | Up to 2 month
  Change in number of lesions detected on MRI during treatment.
Change in NIH Stroke Scale (NIHSS) score | Up to 2 month
  Change in NIH Stroke Scale (NIHSS) score during treatment (comparing scores at 2 weeks post-final dose with baseline scores at initial treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided